CLINICAL TRIAL: NCT04731649
Title: Families Talking Together Plus (FTT+): An Online, Family-Based Approach to Promote Sexual Delay and Strengthen the Evidence-Base for Sexual Risk Avoidance Education
Brief Title: Families Talking Together Plus: An Approach to Promote Sexual Delay and Strengthen Sexual Risk Avoidance Education
Acronym: FTT+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00426772; 90SR0113-01-00 (Other Grant/Funding Number: Administration of Children and Families); PRO00108607 (Other: Duke)
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Families Talking Together; Adolescent Sexual Health; Community Health Workers; Prevention
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sex Education + Standard Care (Experimental): The experimental arm will receive the FTT + intervention
  Interventions: Behavioral: Families Talking Together Plus (FTT +)
- No Education + Standard Care (No Intervention): The control arm will not receive the FTT + intervention

INTERVENTIONS:
Behavioral: Families Talking Together Plus (FTT +) — FTT + consists of three online intervention sessions of approximately 60-90 minutes each, that cover content from nine modules designed to teach parents effective communication skills, build parent-adolescent relationships, help parents develop successful monitoring strategies, and teach adolescents assertiveness, refusal skills, and how to use a condom correctly and every time.
  Arms: Sex Education + Standard Care

SUMMARY:
Despite reductions in adolescent sexual behavior over the past decade, premature sexual activity remains prevalent among adolescents and alarming adolescent sexual and reproductive health (SRH) disparities exist. Positive youth development (PYD) research has identified adolescent protective factors, such as success sequencing, self-regulation, goal setting, and strong family support [i.e., positive family development (PFD)] that are associated with increased sexual risk avoidance as well as individual life opportunities and societal benefits. Needed are programmatic efforts to strengthen adolescent protective factors among populations in greatest need, with a particular emphasis on the important role of parents in promoting sexual delay. The proposed project is designed to target Latino and Black adolescents aged 12-17 years residing in the South Bronx, New York City, a high-need community for sexual risk programming and promotion of adolescent life opportunities. The investigators evaluate a program called Families Talking Together Plus (FTT+), an online, parent-based intervention that is medically accurate, culturally tailored, and age-appropriate. To implement FTT +, the investigators draw upon an innovative and culturally competent intervention delivery approach, namely community health workers (CHWs) as "Life Opportunity Coaches."

DETAILED DESCRIPTION:
Despite reductions in adolescent sexual behavior over the past decade, premature sexual activity remains prevalent among adolescents and alarming adolescent sexual and reproductive health (SRH) disparities exist. The adverse short and long-term consequences of premature adolescent sexual behavior are well-documented, including negative effects on the physical, emotional, social, and economic well-being of youth. Positive youth development (PYD) research has identified adolescent protective factors, such as success sequencing, self-regulation, goal setting, and strong family support [i.e., positive family development (PFD)] that are associated with increased sexual risk avoidance as well as individual life opportunities and societal benefits.

Families Talking Together Plus (FTT +) is an online intervention designed to reduce adolescent sexual risk behavior through supporting caregiver-adolescent communication about sex. The goals of the program are to (1) delay sexual debut, (2) reduce sexual behavior, (3) increase correct and consistent condom use, and (4) increase engagement with community resources among Black and Latino adolescents aged 12-17 years (n=600) residing in a community with disparate adolescent SRH outcomes and high need for improved adolescent life opportunities and success sequencing support, the South Bronx, New York City.

The 2-arm parallel randomized controlled trial (RCT) will evaluate the efficacy of the FTT + intervention in delaying sexual debut, reducing adolescent sexual behavior, and linking adolescents to community resources and services for sexual risk behavior, PYD, and success sequencing. The investigators will recruit adolescents and the primary adult caregivers in the homes using area sampling methods piloted-tested by Center for Latino Adolescent and Family Health (CLAFH) staff with excellent results in our previous research in the target community. Parents and adolescents will complete a questionnaire (separately) at baseline assessments. Subsequently, parent-adolescent dyads will be randomly assigned to either, (1) the experimental group (who will receive the FTT + intervention), or (2) the control group that does not receive any intervention. The baseline sample size will be 600 dyads, with 300 dyads in each group.

Parents randomized to the experimental condition will receive three 60 to 90 minute virtual intervention sessions consisting of 9 modules delivered to the parent by community healthcare workers. Intervention sessions should happen within the first month following the baseline interview. FTT + modules address self-regulation, success sequencing, the benefits of delaying sex, correctly using a condom every time, healthy relationships, goal setting, resisting sexual coercion, dating violence, and other youth risk behaviors such as underage drinking or illicit drug use. In addition, parents receive guidance on effective adolescent monitoring and supervision and strengthening the relationship quality with the adolescent.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between the ages of 12 and 17 years old
* Adolescent must identify as Latino or Black
* Adolescent has a primary caregiver
* Residence in Mott Haven, South Bronx

Exclusion Criteria:

* Adolescent is not between the ages of 12-17
* Adolescent is not Latino or Black
* Adolescent does not have a primary caregiver
* Non-resident of Mott Haven, South Bronx

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1227 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Sexual Debut/Ever Sex (Vaginal) | 9-month post-intervention
  Defined as adolescent report of having engaged in vaginal sex.
Sexual Debut/Ever Sex (Anal) | 9-month post-intervention
  Defined as adolescent report of having engaged in anal sex.
Sexual Debut/Ever Sex (Oral) | 9-month post-intervention
  Defined as adolescent report of having engaged in oral sex.

SECONDARY OUTCOMES:
Frequency of Vaginal Sex Acts | 9-month post-intervention
  Defined as number of vaginal sex acts within a 6-month period
Frequency of Anal Sex Acts | 9-month post-intervention
  Defined as number of anal sex acts within a 6-month period
Frequency of Oral Sex Acts | 9-month post-intervention
  Defined as number of oral sex acts within a 6-month period
Number of Sexual Partners | 9-month post-intervention
  Defined as the number of different sexual partners within a 6-month period
Adolescent Consistency of Condom Use: As Measured by the Condom Use Among Hispanics Scale | 9-month post-intervention
  Defined as frequency of adolescent condom use during vaginal, anal, and oral sex acts, with higher scores indicating greater consistency of condom use [Minimum Score= 0% - indicates that no condom was used during any type of sex act in the past 6 months, Maximum Score= 100% - indicates that a new condom was used for every sex act in the past 6 months.
Uptake of Sexually Transmitted Infection (STI) Testing | 9-month post-intervention
  Defined as adolescent report of utilizing STI testing.
Adolescent Linkage to Community and Healthcare Services: As Measured using the Utilization of Community Resources Scale | 9-month post-intervention
  Measured using the Utilization of Community Resources Scale, with higher scores indicating greater linkage to to services in the community addressing current needs (e.g., food insecurity) & economic capital (e.g., job training) [Minimum score = 0 - indicates no linkage to any services listed; Maximum score= 12- indicates linkage to all types of services listed in scale].
Sexual Debut/Ever Sex (Vaginal) | 3-month post-intervention
  Defined as adolescent report of having engaged in vaginal sex.
Sexual Debut/Ever Sex (Anal) | 3-month post-intervention
  Defined as adolescent report of having engaged in anal sex.
Sexual Debut/Ever Sex (Oral) | 3-month post-intervention
  Defined as adolescent report of having engaged in oral sex.
Frequency of Vaginal Sex Acts | 3-month post-intervention
  Defined as number of vaginal sex acts within a 3-month period
Frequency of Anal Sex Acts | 3-month post-intervention
  Defined as number of anal sex acts within a 3-month period
Frequency of Oral Sex Acts | 3-month post-intervention
  Defined as number of oral sex acts within a 3-month period
Number of Sexual Partners | 3-month post-intervention
  Defined as the number of different sexual partners within a 3-month period
Adolescent Consistency of Condom Use: As Measured by the Condom Use Among Hispanics Scale | 3-month post-intervention
  Defined as frequency of adolescent condom use during vaginal, anal, and oral sex acts, with higher scores indicating greater consistency of condom use [Minimum Score= 0% - indicating no condom use during any type of sex act in the past 3 months, Maximum Score= 100% - indicating condom use for every sex act in the past 3 months.
Uptake of STI Testing | 3-month post-intervention
  Defined as adolescent report of utilizing STI testing.
Adolescent Linkage to Community and Healthcare Services: As Measured using the Utilization of Community Resources Scale | 3-month post-intervention
  Measured using the Utilization of Community Resources Scale, with higher scores indicating greater linkage to services in the community addressing current needs (e.g., food insecurity) & economic capital (e.g., job training) [.minimum score =0 - indicating no linkage to any services listed; maximum score=12- indicating linkage to all types of services listed in scale].

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guilamo-Ramos, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guilamo-Ramos V, Benzekri A, Thimm-Kaiser M. Evaluating the efficacy of an online, family-based intervention to promote adolescent sexual health: a study protocol for a randomized controlled trial. Trials. 2023 Mar 11;24(1):181. doi: 10.1186/s13063-023-07205-3. PMID 36906589
- See also: Study Protocol — https://link.springer.com/article/10.1186/s13063-023-07205-3

DOCUMENTS (1):
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04731649/ICF_000.pdf